CLINICAL TRIAL: NCT00974493
Title: Randomized Open Label Study of Oral Versus Intravenous Antibiotic Treatment for Bone and Joint Infections Requiring Prolonged Antibiotic Treatment: Multi-centre Study
Brief Title: Oral Versus Intravenous Antibiotics for Bone and Joint Infections (OVIVA B&J)
Acronym: OVIVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Matthew Scarborough, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OVIVA
Record Dates: First submitted 2009-09-04; First posted 2009-09-10 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Bone Infection; Joint Infection
Keywords: oral; intravenous; antibiotics; bone; joint; infection
MeSH Terms: conditions — Infections | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral antibiotics (Active Comparator)
  Interventions: Drug: Antibiotics
- Intravenous antibiotics (Active Comparator)
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Antibiotics — The trial protocol does not specify individual antibiotics, as the trial question is one of strategy (i.e. oral vs intravenous route) rather than individual antibiotics.
  Within allocated strategy (i.e. oral or intravenous) antibiotics will be selected by a clinician with reference to the subject's clinical condition, microbiological data and local guidelines.
  Other Names: Individual antibiotics not specified by protocol

SUMMARY:
The study will compare the outcomes of treating bone and joint infections with 6 weeks of intravenous antibiotics with 6 weeks of oral antibiotic treatment. The trial is of antibiotic "strategy" rather than of individual antibiotics. The study will be open label, but the primary outcome will be proven failure of infection treatment, determined by pre-established objective criteria for treatment failure. The null hypothesis tested is that there will be no difference in treatment failure rates.

DETAILED DESCRIPTION:
A long course of antibiotic therapy given by a "drip" (i.e. intravenous) is recommended treatment for many serious bacterial infections. It is costly and inconvenient for the patient to remain hospitalised for therapy, so outpatient antibiotic therapy (OPAT) programmes have been established in many countries to deliver intravenous antibiotics safely and conveniently. The majority of patients referred to OPAT programmes have bone and joint infections. However, there is no clear evidence that bone and joint infection really require long courses of intravenous antibiotics rather than oral antibiotics.

We will compare the outcome of treatment with intravenous versus oral antibiotic therapy for patients with bone and joint infection. The choice of antibiotic is complex, and antibiotics that are suitable oral choices are often not suitable intravenous choices and vice versa. Subjects will therefore be randomized to an oral or intravenous "strategy," rather than to individual antibiotics. Outcomes will be determined by pre-established objective criteria for treatment failure.

We have conducted a pilot study in one centre (Oxford), recruiting approximately 200 patients, and are now expanding to include multi-centre recruitment in the UK, aiming to recruit 1050 patients.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to give informed consent for participation in the study. Has a bone and joint infection one of the following categories;

  1. Native osteomyelitis.
  2. Native joint septic arthritis.
  3. Diabetic foot infection with osteomyelitis.
  4. Prosthetic joint associated infection.
  5. Discitis/ spinal osteomyelitis/ epidural abscess
* Has had at least 48 hours, but not more than 7 days, of IV antibiotic therapy already given after definitive surgical management.
* Has a clinical diagnosis of bacterial infection (caused by any organism excepting mycobacteria).
* Is clinically stable in the opinion of the study clinicians, has no further interventions to treat acute infection required or planned.

Exclusion Criteria:

* Has Staph aureus bacteraemia.
* Has suspected bacterial endocarditis.
* Has suspected mediastinal infection.
* Has suspected central nervous system infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1054 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bejon, PhD, Principal Investigator — Oxford Radcliffe Hospitals Trust; Matthew Scarborough, MB BS, Principal Investigator — Oxford University Hospitals
Locations (2):
- United Kingdom (2):
  - Nuffield Orthopaedic Centre, Oxford, Oxfordshire
  - Oxford Radcliffe Hospitals Trust, Oxford, Oxfordshire

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Antibiotics | Intravenous Antibiotics
Started | 527 | 527
Completed | 509 | 506
Not Completed | 18 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Antibiotics | Intravenous Antibiotics | Total
Number analyzed (Participants) | 527 | 527 | 1054
Age, Customized [Median (Full Range); unit: years] | 60 [18 to 91] | 61 [18 to 92] | 60 [18 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 207 | 376
  Male | 358 | 320 | 678
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 527 | 527 | 1054

OUTCOME MEASURES:

1. Primary Outcome: The Frequency of Definite Failure of Infection Treatment.
Description: Number of participants with definite failure of infection treatment defined by microbiological, histological and clinical criteria and assessed by an independent blinded endpoint committee
Time Frame: 1 year
Population: Modified ITT (excluding participants without available endpoint data)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Antibiotics | Intravenous Antibiotics
Number analyzed (Participants) | 509 | 506
Participants | 67 | 74

ADVERSE EVENTS:
Arm/Group | Oral Antibiotics | Intravenous Antibiotics
All-Cause Mortality (participants affected / at risk) | 6/527 | 17/527
Serious Adverse Events (participants affected / at risk) | 138/527 | 146/527
Other Adverse Events (participants affected / at risk) | 80/527 | 86/527
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Oral Antibiotics (N=527) | Intravenous Antibiotics (N=527)
All (General disorders) | 138 | 146 — Adverse Event data were not available for 8 participants in relation to C difficile and Line Complication. For events collected by non-systematic methods, data are reported with reference to organ system rather than specific adverse event term
C difficile (Infections and infestations) | 5/523 | 9/523 — C difficile was reported as a defined secondary outcome. No data available from 4 participants in each arm
Line complication (Injury, poisoning and procedural complications) | 5/523 | 49/523 — Line complications were reported as a defined secondary outcome. No data available from 4 participants in each arm
Neurological (Nervous system disorders) | 10 | 4
Cardiovascular (Cardiac disorders) | 29 | 26
Respiratory (Respiratory, thoracic and mediastinal disorders) | 21 | 14
Gastrointestinal (Gastrointestinal disorders) | 13 | 21
Renal (Renal and urinary disorders) | 12 | 11
Diabetic (Endocrine disorders) | 10 | 7
Neoplastic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 21 | 17
Skin and soft tissue unrelated to original surgical site (Skin and subcutaneous tissue disorders) | 7 | 10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Antibiotics (N=527) | Intravenous Antibiotics (N=527)
Related to the operative site (General disorders) | 69 | 46 — Includes directed specialist care for symptom control, wound management, mobility, skin and soft tissue infection, dislocation or recurrent primary endpoint
Antibiotic related (General disorders) | 15 | 30 — Antibiotic related events represented here were attributed by the responsible infection specialist to antibiotic therapy (as opposed to unrelated co-morbidities).
Frailty related (General disorders) | 5 | 10 — Frailty related events included slips, trips or falls in the elderly or readmission as a result of inability to cope at home

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No